CLINICAL TRIAL: NCT00253721
Title: Intra-Arterial Melphalan (L-Phenylalanine Mustard) Administered in Conjunction With Osmotic Blood-Brain Barrier Disruption in Patients With Brain Malignancies: A Phase I Study
Brief Title: Melphalan With BBBD in Treating Patients With Brain Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Other competing clinical trials affecting enrollment
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00001299; P30CA069533 (NIH); 1299 (Other: OHSU eIRB); ONC-98018-L (Other: OHSU Knight Cancer Institute); 4834 (Other: OHSU IRB (discontinued number))
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma; Metastatic Cancer
Keywords: adult anaplastic astrocytoma; adult brain stem glioma; adult diffuse astrocytoma; adult central nervous system germ cell tumor; adult medulloblastoma; adult supratentorial primitive neuroectodermal tumor (PNET); adult anaplastic oligodendroglioma; adult oligodendroglioma; adult pineoblastoma; tumors metastatic to brain; adult mixed glioma; recurrent adult brain tumor; primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma; Neoplasm Metastasis; Astrocytoma; Medulloblastoma; Oligodendroglioma; Pinealoma; Brain Neoplasms; Glioma | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects (Experimental)
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Melphalan — All levels: Every 4 weeks for up to one year
  Dose Escalation Plan:
  Level 1: 4mg/m2/day x 2 days
  Level 2: 6mg/m2/day x 2 days
  Level 3: 8mg/m2/day x 2 days
  Level 4: 10mg/m2/day x 2 days
  Level 5: 12mg/m2/day x 2 days

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving drugs directly into the arteries around the tumor may kill more tumor cells. Mannitol may open the blood vessels around the brain [Blood-Brain Barrier Disruption (BBBD)]and allow melphalan to be carried directly to the brain tumor. Giving melphalan together with BBBD may be an effective treatment for central nervous system cancer.

PURPOSE: This phase I trial is studying side effects and best dose of melphalan when given together with mannitol in treating patients with central nervous system cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of intra-arterial melphalan when given in combination with BBBD in patients with primary or metastatic central nervous system (CNS) malignancy.
* Determine the toxic effects of melphalan given with BBBD in these patients.
* Determine, preliminarily, the efficacy of this regimen in these patients.

OUTLINE: This is a dose-escalation study of melphalan.

Patients receive intra-arterial mannitol with BBBD followed by intra-arterial melphalan over 10 minutes on days 1 and 2*. Treatment repeats every 4 weeks for up to 12 monthly courses in the absence of disease progression or unacceptable toxicity .

NOTE: *Patients with gliomas localized to the posterior circulation (i.e., brain stem gliomas) receive melphalan on day 1 only.

Cohorts of 3-6 patients receive escalating doses of melphalan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study therapy, patients are followed every 3 months for 1 year; every 6 months for the next 2 years; then annually.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Signed written informed consent form in accordance with institutional guidelines
* Histologically confirmed primary or metastatic CNS malignancy (Patients with metastatic disease must have histological confirmation of the primary cancer AND confirmation by surgical specimen, cerebrospinal fluid cytology, elevated tumor markers, or clinical evidence of CNS involvement)
* Single or multiple cerebellar or cerebral cortex lesions allowed
* Life expectancy at least 60 days
* Radiographically evaluable disease by MRI or CT scan
* Age 18 years or older
* At least 28 days since prior radiotherapy (systemic, cranial, and/or spinal)
* At least 28 days since prior chemotherapy (42 days for nitrosoureas)
* Adequate cardiac and pulmonary function to tolerate general anesthesia
* Performance status of Eastern Cooperative Oncology Group (ECOG) 0-2
* Other tumor masses in the spinal cord allowed provided there is no radiographic or clinical evidence of spinal cord block
* Available for follow-up for at least one year following completion of treatment
* Fertile patients must use effective contraception for 2 months prior to, during, and for 3 months after study participation
* Pre-treatment lab tests within 14 days prior to initiation of treatment:

  * White blood cell count (WBC) > 2,500/mm^3
  * Absolute granulocyte count > 1,200/mm^3
  * Platelet count > 100,000/mm^3
  * Hematocrit > 30% (transfusion allowed)
  * Bilirubin ≤ 2 times upper limit of normal (ULN)
  * Serum glutamic oxaloacetic transaminase (SGOT) ≤ 3 times ULN
  * Creatinine ≤ 2 times ULN
* Subjects with history of smoking or emphysema require diffusing capacity of lung for carbon monoxide (DLCO) ≥ 80% of predicted value for age
* Histological sections submitted for pathology review

EXCLUSION CRITERIA:

* Radiographic evidence of excessive intra-cranial mass effect and/or spinal block
* Known hypersensitivity or intolerance to melphalan
* NCI CTC Grade 3 or greater baseline neurologic symptoms
* Immunologically compromised (Concurrent corticosteroids for tumor edema allowed)
* Unable to tolerate general anesthesia
* Pregnant, positive human chorionic gonadotropin (HCG) test, or lactating
* HIV positive
* Receiving concurrent radiotherapy or immunotherapy
* Serious illness that would preclude study participation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 1998-05; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD)of Melphalan as measured by NCI common toxicity criteria (CTC) v2 toxicities | 5 years
  MTD = dose of Melphalan that produces grade 3 neurotoxicity in 33% of subjects

SECONDARY OUTCOMES:
Efficacy of chemotherapy regimen as measured by clinical and radiographic response from first day of treatment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward A. Neuwelt, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon, United States